CLINICAL TRIAL: NCT06193434
Title: A Phase 1 FIH, Randomized, Double Blind, Placebo Controlled, SAD/MAD Study to Assess Safety, Tolerability and PK in Healthy Participants and in Atopic Dermatitis Patients
Brief Title: A First In Human (FIH) Study of IBI356 in Healthy Participants and in Atopic Dermatitis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIBI356A101CN
Record Dates: First submitted 2023-12-12; First posted 2024-01-05 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants; Atopic Dermatitis Patients
MeSH Terms: interventions — mycophenolic adenine dinucleotide; dupilumab; Sagittal Abdominal Diameter

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- IBI356 for Single ascending dose (SAD) (Experimental)
  Interventions: Drug: IBI356 for SAD
- IBI356 for Multiple ascending dose (MAD) (Experimental)
  Interventions: Drug: IBI356 for MAD
- Placebo for MAD (Placebo Comparator)
  Interventions: Drug: Placebo for MAD
- Dupilumab for MAD (Active Comparator)
  Interventions: Drug: Dupilumab for MAD
- Placebo for SAD (Placebo Comparator)
  Interventions: Drug: Placebo for SAD

INTERVENTIONS:
Drug: IBI356 for MAD — Receive IBI356 in a multiple dose.
  Arms: IBI356 for Multiple ascending dose (MAD)
Drug: Dupilumab for MAD — Active comparator
  Arms: Dupilumab for MAD
Drug: IBI356 for SAD — Receive IBI356 in a single dose.
  Arms: IBI356 for Single ascending dose (SAD)
Drug: Placebo for SAD — Receive placebo in a single dose.
  Arms: Placebo for SAD
Drug: Placebo for MAD — Receive placebo in a multiple dose.
  Arms: Placebo for MAD

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of IBI356 in Healthy Participants and in Atopic Dermatitis Patients

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants:

   1. Aged 18 to 45 years,
   2. Weight 50 to 120 kgs,
   3. Good physical and mental health based on medical history, physical examination, clinical laboratory, ECG, and vital signs, as judged by the Investigator.
   4. No child-bearing potential during the trial and within 6 months after SAD doses, and adequate contraceptive measures can be taken.
2. Atopic dermatitis:

   1. Aged 18 to 75 years,
   2. body mass index (BMI): 18.0 - 32.0 kg/m2,
   3. Atopic Dermatitis (AD) for 1 year or longer at Baseline,
   4. Eczema Area and Severity Index (EASI) of 16 or higher at baseline,
   5. Investigator Global Assessment (IGA) of 3 or 4 at baseline,
   6. AD involvement of 10 percent or more of body surface area at Baseline,
   7. Documented history, within 1 year before Baseline, of either inadequate response to topical treatments or inadvisability of topical treatments,
   8. Must have applied a stable dose of topical bland emollient at least twice daily for at least 7 consecutive days before Baseline.

Exclusion Criteria:

1. History of relevant drug allergies.
2. Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (for example, compromise the well-being) of the participant or that could prevent, limit, or confound the protocol-specified assessments
3. Healthy participants:

   1. History of alcohol abuse or drug addiction within 1 year before screen,
   2. Positive drug and alcohol screen at screening.
4. Atopic dermatitis:

   1. Having used any of the following treatments within 4 weeks before the baseline visit, or any condition that, in the opinion of the investigator, was likely to require Immunosuppressive/ immunomodulating drugs treatment(s) during the first 4 weeks of study treatment:
   2. Treatment with topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) within 1 week before the baseline visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Event (AE) in SAD study. | Baseline to Week 20
Occurrence of Adverse Event (AE) in MAD study. | Baseline to Week 36
Occurrence of Serious Adverse Event (SAE) in SAD study. | Baseline to Week 20
Occurrence of Serious Adverse Event (SAE) in MAD study. | Baseline to Week 36
Changes in blood pressure mmHg (as a measure of safety and tolerability) in SAD study. | Baseline to Week 20
Changes in blood pressure mmHg (as a measure of safety and tolerability) in MAD study. | Baseline to Week 36
Changes in respiratory rate measured as breaths per minute (as a measure of safety and tolerability) in SAD study. | Baseline to Week 20
Changes in respiratory rate measured as breaths per minute (as a measure of safety and tolerability) in MAD study. | Baseline to Week 36
Changes in heart rate bpm (as a measure of safety and tolerability) in SAD study. | Baseline to Week 20
Changes in heart rate bpm (as a measure of safety and tolerability) in MAD study. | Baseline to Week 36
Changes in tympanic temperature °C in SAD study. | Baseline to Week 20
Changes in tympanic temperature °C in MAD study. | Baseline to Week 36
Changes in electrocardiograms PR, QR, QRS and QT intervals (as a measure of safety and tolerability) in SAD study. | Baseline to Week 20
Changes in electrocardiograms PR, QR, QRS and QT intervals (as a measure of safety and tolerability) in MAD study. | Baseline to Week 36

SECONDARY OUTCOMES:
Area under the concentration time curve from time 0 to last observation (AUC 0-t). | Baseline to Week 16
Maximum observed concentration (Cmax) after infusion. | Baseline to Week 16
Systemic clearance after infusion (CL). | Baseline to Week 16
Volume of distribution during the terminal phase after infusion(Apparent volume of distribution, V). | Baseline to Week 16
Elimination half-life during the terminal phase after infusion(Half-life, t1/2). | Baseline to Week 16
To assess immunogenicity: production of anti-drug antibodies (ADA) following SAD and Multiple ascending dose(MAD) doses. | Baseline to Week 16

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No